CLINICAL TRIAL: NCT06763276
Title: The Effect of Preoperative Virtual Reality Cartoon Viewing on Postoperative Pain and Anxiety in Children Undergoing Tonsillectomy and Adenoidectomy
Brief Title: Preoperative VR Cartoon Viewing Reduces Postoperative Pain and Anxiety in Pediatric Tonsillectomy Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Tinaztepe University (Other)
Responsible Party: Principal Investigator, Berna Dizer, Assistant professor, Izmir Tinaztepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İzmirTınaztepeÜ-B.Dizer-001
Record Dates: First submitted 2024-07-26; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Tonsillectomy; Adenoidectomy
Keywords: Virtual Reality; Cartoon; Pain Level; Anxiety Level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): A meeting was conducted with the children and their parents. Information about the content of the research was provided. Consent forms were completed by the children and their parents. Instructions on how to use the virtual reality headset were given to the children and their parents.
  Mothers were asked to comfort and caress their children during the preoperative period.
  The first 15-20 minutes of the cartoon were shown to the children before the surgery. After watching the cartoon, the children were sent for tonsillectomy and adenoidectomy surgery. The remainder of the cartoon was shown one hour after the surgery once the child had settled in the recovery room.
  Before the tonsillectomy and adenoidectomy surgery, immediately after the child returned to the ward post-surgery, and 8 hours after the surgery:
  The child's vital signs were recorded. The child's anxiety and pain scores were assessed.
  Interventions: Other: Virtual Reality Group
- Control Group (No Intervention): Consent forms were completed by the children and their parents. Mothers were asked to comfort and caress their children.
  Before the tonsillectomy and adenoidectomy surgery, immediately after the child returned to the ward post-surgery, and 8 hours after the surgery:
  The child's vital signs were recorded. The child's anxiety and pain scores were assessed. The children in the control group were allowed to watch the cartoon via virtual reality (VR) after all data for the research had been collected to ensure ethical equality.

INTERVENTIONS:
Other: Virtual Reality Group — In the study, a 400-gram virtual reality (VR) headset with an anti-reflective lens system was used, compatible with all earphones with screens ranging from 4.5 to 7.0 inches. The virtual reality (VR) headset, which was lightweight enough for children to wear, was supported on three sides to fit securely on the children's heads and was disinfected after each use. For the experimental group, the compartment at the front of the virtual reality (VR) headset was removed. The earphone was placed into the removed compartment, which was then reinserted. Subsequently, the YouTube virtual reality (VR) feature was activated on the phone, making it ready for viewing.
  Arms: Virtual Reality Group

SUMMARY:
The aim of this study is to determine the effect of watching a cartoon with a virtual reality headset before surgery on the pain and anxiety levels of children aged 7-12 years.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of watching a cartoon with a virtual reality headset before surgery on the pain and anxiety levels of children aged 7-12 years. In line with this aim, children aged 7-12 who were scheduled for tonsillectomy and adenoidectomy at the Ear, Nose, and Throat Department of Uşak University Education and Research Hospital were shown a cartoon with a virtual reality headset before surgery, and their pain and anxiety levels were examined. The study was conducted as a randomized controlled experimental study at the Ear, Nose, and Throat Unit of Uşak University Education and Research Hospital. The population of the study consisted of children aged 7-12 who applied for tonsillectomy and adenoidectomy surgery at the Ear, Nose, and Throat Unit of Uşak University Education and Research Hospital. The sample of the study included a total of 102 children, with 51 in the experimental group and 51 in the control group, who met the research criteria and volunteered to participate in the study between November 10, 2023, and June 1, 2024. Data collection tools included the informed consent form, sociodemographic questionnaire, vital signs assessment form, Visual Analog Scale, and the Perioperative Multidimensional Anxiety Scale for children.

ELIGIBILITY:
Inclusion Criteria:

Child's criteria:

* Children aged between 7 and 12 years
* Ability to understand pain and anxiety scales
* Possession of communication skills
* Absence of mental issues
* Absence of physical illnesses
* Absence of chronic illnesses
* Willingness of the child and family to participate in the study
* No visual, hearing, or speech problems

Exclusion Criteria:

* Children younger than 7 years or older than 12 years
* Presence of any chronic illness that could affect pain and anxiety levels
* Presence of psychosocial issues
* Children or parents who meet the inclusion criteria but do not wish to wear the virtual reality headset (VRH) glasses
* Children who need to wear glasses other than the virtual reality headset (VRH)
* Children with hearing problems
* Children who do not wish to watch the shrek cartoon

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
Vital signs | Preoperative, immediately postoperative, and 8 hours postoperative.
  Systolic Blood Pressure (mmHg) Description: Systolic blood pressure levels measured during the perioperative period.
Diastolic Blood Pressure (mmHg) | Preoperative, immediately postoperative, and 8 hours postoperative
  Diastolic blood pressure levels will be measured to assess changes in blood pressure during the perioperative period.
Heart Rate (bpm) | Preoperative, immediately postoperative, and 8 hours postoperative
  Heart rate will be measured to monitor cardiac activity during the perioperative period.
Body Temperature (°C) | Preoperative, immediately postoperative, and 8 hours postoperative
  Body temperature will be measured to observe temperature changes during the perioperative period.
Hemoglobin (g/dL) | Preoperative and 24 hours postoperative
  Hemoglobin levels will be measured preoperatively and within 24 hours postoperatively to evaluate changes in blood parameters during the perioperative period.
Creatinine (mg/dL) | Preoperative and 24 hours postoperative
  Creatinine levels will be measured preoperatively and within 24 hours postoperatively to monitor renal function during the perioperative period.
Glucose (mg/dL) | Preoperative and 24 hours postoperative
  Glucose levels will be measured preoperatively and within 24 hours postoperatively to assess perioperative glucose regulation

SECONDARY OUTCOMES:
Secondary Outcome Measure | Preoperative, immediately postoperative, 8 hours postoperative
  Pain Score: The Visual Analog Scale (VAS) was used to measure pain intensity in children during the postoperative period following tonsillectomy and adenoidectomy. The children were assessed using the Visual Analog Scale (VAS) before surgery, immediately after returning to the ward post-surgery, and 8 hours after surgery.The Visual Analog Scale (VAS) ranges from 0 to 10, with 0 indicating no pain and 10 representing the worst possible pain. Higher scores indicate greater pain intensity.

OTHER OUTCOMES:
Tertiary Outcome Measure | Preoperative, immediately postoperative, 8 hours postoperative
  Anxiety Score: The Perioperative Multidimensional Anxiety Scale for Children is a visual analog scale consisting of 5 items, each scored between 0 and 100. The scale was used to measure anxiety levels in children during the perioperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Tinaztepe University, Izmir, Buca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mersin SK, Dizer B, Tuna A. Effect of preoperative virtual reality cartoon viewing on postoperative pain and anxiety in children undergoing tonsillectomy and adenoidectomy: A randomized controlled trial. PLoS One. 2025 Sep 11;20(9):e0331793. doi: 10.1371/journal.pone.0331793. eCollection 2025. PMID 40934240